CLINICAL TRIAL: NCT05307315
Title: The Effect of Listening to Music Before Surgery on the Anxiety of Individuals Scheduled for Urological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZBU-SBE-NESLİHAN-AKER-0000-85
Record Dates: First submitted 2021-10-19; First posted 2022-04-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2021-10

CONDITIONS: Preoperative Anxiety
Keywords: preoperative anxiety; surgery anxiety; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music (Experimental): The state/trait anxiety inventory and surgery-specific anxiety inventory will be administered to the experimental group before the surgery. Then they will listen to Turkish Classical Music for 30 minutes.
  The scales will be applied again 15 minutes after the music ends.
  Interventions: Other: listening to music
- control (No Intervention): The state/trait anxiety inventory and surgery-specific anxiety scale will be administered to the control group before surgery. The same scales will be applied again 45 minutes after the scales are applied.

INTERVENTIONS:
Other: listening to music — The experimental group will listen to Turkish instrumental music with headphones for 30 minutes.
  Other Names: music
  Arms: music

SUMMARY:
Many patients before the operation feel a high level of anxiety. This felt anxiety can develop due to many reasons such as anesthesia, not being able to wake up from the surgery and being disabled, and fear of feeling pain after the surgery. Music applications, which are among non-pharmacological techniques, are frequently used in the management of pain and anxiety.In this study, the effect of listening to music in the preoperative period on the anxiety of urology patients will be investigated

DETAILED DESCRIPTION:
The anxiety felt at a high level in many patients in the pre-operative period can be caused by many reasons such as general anesthesia, anxiety about not being able to wake up from the operation, fear of being disabled, fear of pain after the operation, fear of losing control over the body, fear of sexual loss and worries about not being able to work after the operation can develop. Anxiety experienced at a high level in the preoperative period; While it causes physical problems such as dizziness, nausea and headache, it also affects the anxiety to be experienced after the surgery. Looking at the effects of preoperative anxiety in the postoperative period, it increases the intensity of postoperative pain and analgesia requirement, affects anesthesia requirements, and increases hospitalization time in some types of surgery, and as a result, increases postoperative morbidity and mortality. Anxiety levels of patients; may be affected by a wide variety of factors such as previous experiences, the way they came to the hospital, their gender, age, and the type of surgery they will undergo. In contrast, effective control of preoperative anxiety provides better management of postoperative pain and faster recovery.

The positive and curative effect of music has been the subject of constant interest from past to present and it has been used more and more among non-pharmacological techniques. Listening to music, intensive care, surgery, psychiatry, obstetrics, pediatrics, oncology services, in the process of radiotherapy and chemotherapy in patients with other diagnostic and treatment from the symptoms that arise in the process, especially in the management of pain and anxiety is often applied. In addition, it has been determined that it has important positive effects on the activation of the immune system, increasing the quality of life, reducing the amount of drugs used in the treatment of pain, shortening the hospital stay and spirituality.

In many studies in the literature examining the effect of music on anxiety associated with surgical intervention; it has been found that music reduces the level of anxiety. However, a study has also found that music does not affect the anxiety experienced by an individual. Although there are no studies evaluating the effect of music on the anxiety level of individuals scheduled for urological surgery, in a meta-analysis study evaluating the effect of music on individuals undergoing urological procedures in outpatients, it was found that music reduces anxiety.

In the nursing profession, which focuses on providing holistic care in the biopsychosocial sense, it is important to increase the quality of care by addressing the emotional experiences of the individual during physical health problems.Addressing anxiety as an emotional experience before surgical intervention within the scope of nursing interventions may contribute to increasing the quality of life of the individual.In the light of this information, this study aims to evaluate the effect of listening to music before surgery on the anxiety level of individuals who are planned for urological surgery as an independent therapeutic nursing intervention and to improve nursing care with the findings obtained from the study.

ELIGIBILITY:
Inclusion Criteria:

* To be literate
* Being undergoing urological surgery for the first time
* Be over 18 years old
* Having agreed to participate in the study

Exclusion Criteria:

* To be hard of hearing
* Inability to communicate verbally
* Having a disease that prevents data collection
* Having difficulty wearing headphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Measuring the preoperative anxiety level of the experimental group with the State-Trait Anxiety Inventory | within 5 hours before surgery
  The preoperative anxiety levels of the experimental group will be measured with the State-Trait Anxiety Inventory. Scores from the scale range from 20 to 80. High scores indicate a high level of anxiety.
Measuring the preoperative anxiety level of the control group with the State-Trait Anxiety Inventory | within 5 hours before surgery
  The preoperative anxiety levels of the control group will be measured with the State-Trait Anxiety Inventory. Scores from the scale range from 20 to 80. High scores indicate high levels of anxiety.
Measuring the preoperative anxiety level of the experimental group with the State-Trait Anxiety Inventory after listening to music for 30 minutes | 15 minutes after listening to music
  After listening to music for 30 minutes in the experimental group, their preoperative anxiety levels will be measured with the State-Trait Anxiety Inventory. Scores from the scale range from 20 to 80. High scores indicate a high level of anxiety.
Measuring the preoperative anxiety level of the control group without listening to music with the State-Trait Anxiety Inventory | 45 minutes after the first scales are applied
  Preoperative anxiety levels will be measured with the State-Trait Anxiety Inventory, 45 minutes after the first scales are applied, without listening to music in the control group. Scores from the scale range from 20 to 80. High scores indicate a high level of anxiety.

SECONDARY OUTCOMES:
Measuring the preoperative anxiety level of the experimental group with the Surgery-Specific Anxiety Scale | within 5 hours before surgery
  The preoperative anxiety levels of the experimental group will be measured with the Surgery-Specific Anxiety Scale. The maximum score from the scale is 50. High scores indicate a high level of anxiety.
Measuring the preoperative anxiety level of the control group with the Surgery-Specific Anxiety Scale | within 5 hours before surgery
  The preoperative anxiety levels of the control group will be measured with the Surgery-Specific Anxiety Scale. The maximum score that can be obtained from the scale is 50. High scores indicate high levels of anxiety.
Measuring the preoperative anxiety level of the experimental group with the Surgery-Specific Anxiety Scale after listening to music for 30 minutesmusic | 15 minutes after listening to music
  After listening to music for 30 minutes in the experimental group, their preoperative anxiety levels will be measured with the Surgery-Specific Anxiety Scale. The maximum score from the scale is 50. High scores indicate a high level of anxiety.
Measuring the preoperative anxiety level of the control group without listening to music with the Surgery-Specific Anxiety Scale | 45 minutes after the first scales are applied
  Preoperative anxiety levels will be measured with the Surgery-Specific Anxiety Scale, 45 minutes after the first scales are applied, without listening to music in the control group. The maximum score from the scale is 50. High scores indicate a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Arguvanlı Çoban, Study Director — Bülent Ecevit Üniversity; Neslihan Aker, Principal Investigator — Bülent Ecevit Üniversity
Locations (1):
- Neslihan Aker, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared